CLINICAL TRIAL: NCT01399697
Title: A Multi-center Study of the Safety and Effect on Disease Activity of Tocilizumab (TCZ) in Combination With MTX Versus Tocilizumab Monotherapy in Patients With Rheumatoid Arthritis, With Inadequate Response to MTX (Defined as DAS 28 > 3,2)
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Combination With Methotrexate Versus RoActemra/Actemra Monotherapy in Patients With Rheumatoid Arthritis and an Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML27828
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: methotrexate; Drug: tocilizumab [RoActemra/Actemra]
- B (Active Comparator)
  Interventions: Drug: methotrexate; Drug: placebo; Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: methotrexate — orally, Week 1 - 16
Drug: methotrexate — orally, Week 17-28
  Arms: A
Drug: placebo — methotrexate placebo orally, Week 17-28
  Arms: B
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg iv every 4 weeks, 28 weeks

SUMMARY:
This randomized, double-blind, parallel-group study will evaluate the efficacy and safety of RoActemra/Actemra (tocilizumab) in combination with methotrexate versus RoActemra/Actemra monotherapy in patients with rheumatoid arthritis and an inadequate response to methotrexate. All patients will receive RoActemra/Actemra 8 mg/kg intravenously (iv) every 4 weeks plus oral methotrexate for 16 weeks. Patients achieving low disease activity at Week 16 will be randomized to receive a further 12 weeks of RoActemra/Actemra treatment plus either methotrexate or placebo. Anticipated time on study treatment is 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Active moderate to severe rheumatoid arthritis (DAS28 >/= 3.2) at baseline
* Currently receiving methotrexate for at least 12 weeks, at a stable oral dose of at least 15 mg/week for at least 6 weeks prior to treatment (Day 1)
* Body weight < 150 kg
* Oral corticoids must have been at stable dose for at least 25 out of 28 days prior to baseline; maximum dose 10 mg/day

Exclusion Criteria:

* Pregnant or nursing women
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months after baseline
* Rheumatic autoimmune disease other than RA
* Functional class IV as defined by the American College of Rheumatology (ACR) Classification of Functional Status in Rheumatoid Arthritis
* Prior history of or current inflammatory joint disease other than RA
* Treatment with a biologic agent at any time prior to baseline
* Treatment with traditional DMARDs other than methotrexate within 1 month (for leflunomide 3 months) prior to baseline
* Intraarticular or parenteral corticosteroids within 6 weeks prior to baseline
* Previous treatment with RoActemra/Actemra
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Known active current or history of recurrent infection
* History of or currently active primary or secondary immunodeficiency
* Active tuberculosis requiring treatment within the previous 3 years
* Positive for HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- Spain (41):
  - Albacete, Albacete
  - Orihuela, Alicante
  - Torrevieja, Alicante
  - Villajoyosa, Alicante
  - Badajoz, Badajoz
  - Mérida, Badajoz
  - Menorca, Balearic Islands
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Granollers, Barcelona
  - Terrassa, Barcelona
  - Cáceres, Caceres
  - Cadiz, Cadiz
  - Torrelavega, Cantabria
  - Villarreal, Castellon
  - Córdoba, Cordoba
  - Granada, Granada
  - Guadalajara, Guadalajara
  - A Coruña, La Coruña
  - Santiago de Compostela, La Coruña
  - Las Palmas de Gran Canaria, Las Palmas
  - León, Leon
  - Lugo, Lugo
  - Alcalá de Henares, Madrid
  - Fuenlabrada, Madrid
  - Madrid, Madrid
  - Valdemoro, Madrid
  - Málaga, Malaga
  - Cartagena, Murcia
  - El Palmar, Murcia
  - Vigo, Pontevedra
  - Salamanca, Salamanca
  - Seville, Sevilla
  - Santa Cruz de Tenerife, Tenerife
  - Toledo, Toledo
  - Manises, Valencia
  - Valencia, Valencia
  - Valenica, Valencia
  - Barakaldo, Vizcaya
  - Bilbao, Vizcaya
  - Galdakao, Vizcaya

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab (TCZ) Plus (+) Methotrexate (Not Randomized): Participants received TCZ 8 milligrams per kilogram (mg/kg; maximum 800 mg) via intravenous (IV) infusion every 4 weeks (q4w) through Week 24 (total of 7 infusions). Participants also received methotrexate (MTX) capsules orally, at a stable dose (10, 15, 17.5, or 20 mg, no maximum dose was defined) weekly from Week 1 through 16.
- TCZ + MTX (Randomized): Participants received TCZ 8 mg/kg (maximum 800 mg) via IV infusion q4w through Week 24 (total of 7 infusions). Participants also received MTX capsules, orally, at a stable dose (10, 15, 17.5, or 20 mg/week, but no maximum dose was defined), weekly, from Weeks 1 through 24.
- TCZ + Placebo (Randomized): Participants received TCZ 8 mg/kg (maximum 800 mg) via IV infusion q4w through Week 24 (total of 7 infusions). Participants also received MTX capsules, orally, at stable dose (10, 15, 17.5, or 20 mg per week, but no maximum dose was defined) weekly, from Weeks 1 through 16 followed by matching placebo capsules, orally, weekly through Week 24.
Period: Overall Study
Arm/Group | Tocilizumab (TCZ) Plus (+) Methotrexate (Not Randomized) | TCZ + MTX (Randomized) | TCZ + Placebo (Randomized)
Started | 96 | 83 | 82
Completed | 55 | 80 | 78
Not Completed | 41 | 3 | 4
Not completed — Adverse Event | 13 | 3 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0
Not completed — Investigator Decisión | 1 | 0 | 2
Not completed — Lack of Efficacy | 9 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Non-Compliant | 1 | 0 | 0
Not completed — Inclusion Error | 2 | 0 | 0
Not completed — Positive result for hepatitis B | 1 | 0 | 0
Not completed — Clinical RA remission | 1 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated population
Groups:
- TCZ + MTX (Not Randomized): Participants received TCZ 8 mg/kg (maximum 800 mg) via IV infusion q4w through Week 24 (total of 7 infusions). Participants also received MTX capsules orally, at a stable dose (10, 15, 17.5, or 20 mg, no maximum dose was defined) weekly from Week 1 through 16.
- Total: Total of all reporting groups
Arm/Group | TCZ + MTX (Not Randomized) | TCZ + MTX (Randomized) | TCZ + Placebo (Randomized) | Total
Number analyzed (Participants) | 96 | 83 | 82 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (13.2) | 50.2 (12.5) | 51.0 (12.2) | 51.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 62 | 65 | 203
  Male | 20 | 21 | 17 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in Disease Activity Score Based on 28-Joint Count (DAS28) From Week 16 to Week 28
Description: The DAS28 is a combined index for measuring disease activity in rheumatoid arthritis (RA). The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (erythrocyte sedimentation rate [ESR] in millimeters per hour [mm/hr]), and general health status (participant global assessment of disease activity using visual analog scale [VAS], range 1-100 mm). DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Baseline, Week 16, and Week 28
Population: Intent-to-treat (ITT) population: all randomized participants who received at least one dose of study medication and who had at least one efficacy measurement performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- TCZ + MTX (Randomized): TCZ 8 mg/kg (maximum 800 mg) IV q4w along with MTX orally at a stable dose (10, 15, 17.5 or 20 mg/week) up to Week 28.
- TCZ + Placebo (Randomized): TCZ 8 mg/kg (maximum 800 mg) q4w IV up to Week 28 along with MTX orally at stable dose (10, 15, 17.5 or 20 mg per week) up to Week 16 followed by placebo matched to MTX along with TCZ up to Week 28.
Arm/Group | TCZ + MTX (Randomized) | TCZ + Placebo (Randomized)
Number analyzed (Participants) | 83 | 82
units on a scale
  Baseline | 5.42 (1.01) | 5.29 (1.01)
  Week 16 | 1.77 (0.77) | 1.96 (0.76)
  Week 28 | 1.82 (1.18) | 1.98 (1.13)
Statistical Analysis 1: Comparison: TCZ + MTX (Randomized) vs TCZ + Placebo (Randomized); Test type: Superiority or Other; p = 0.700, ANCOVA

2. Secondary Outcome: Percentage of Participants With DAS28 Score Less Than (<) 2.6 at Week 28
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (ESR in mm/hr), and general health status (participant global assessment of disease activity using VAS, range 1-100 mm). DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores indicate worsening. DAS28 <2.6 equals (=) remission.
Time Frame: Week 28
Population: ITT Population; only participants with Week 28 DAS28 values were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TCZ + MTX (Randomized) | TCZ + Placebo (Randomized)
Number analyzed (Participants) | 79 | 79
percentage of participants | 82.3 | 75.9
Statistical Analysis 1: Comparison: TCZ + MTX (Randomized) vs TCZ + Placebo (Randomized); Test type: Superiority or Other; p = 0.328, Chi-squared

3. Secondary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) <2.8 at Week 28
Description: CDAI is the sum of tender and swollen joint count based on 28 joints and the participant and physician global disease assessment (VAS 0-10 centimeters [cm]). CDAI total score 0-76; higher scores = greater affect due to disease activity. CDAI <2.8 = clinical remission.
Time Frame: Week 28
Population: ITT Population; only participants with CDAI scores at Weeks 28 were included in the analysis.
Measure: Number; unit: percentage of participants
Groups:
- Tocilizumab + Methotrexate (Randomized): TCZ 8 mg/kg (maximum 800 mg) IV q4w along with MTX orally at a stable dose (10, 15, 17.5 or 20 mg/week) up to Week 28.
- Tocilizumab + Placebo (Randomized): TCZ 8 mg/kg (maximum 800 mg) q4w IV up to Week 28 along with MTX orally at stable dose (10, 15, 17.5 or 20 mg per week) up to Week 16 followed by placebo matched to MTX along with TCZ up to Week 28.
Arm/Group | Tocilizumab + Methotrexate (Randomized) | Tocilizumab + Placebo (Randomized)
Number analyzed (Participants) | 81 | 81
percentage of participants | 40.7 | 35.8
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate (Randomized) vs Tocilizumab + Placebo (Randomized); Test type: Superiority or Other; p = 0.518, Chi-squared

4. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) <3.3 at Week 28
Description: SDAI is calculated by a simple numerical sum of tender and swollen joint count (based on a 28-joint assessment), participant and physician global assessment of disease activity (VAS 0-10 cm), and level of C-reactive protein in milligram per deciliter (mg/dL). SDAI total score 0-86; higher scores = greater affect due to disease activity. SDAI <3.3 = clinical remission.
Time Frame: 28 weeks
Population: ITT Population; only participants with SDAI scores at Week 28 were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TCZ + MTX (Randomized) | TCZ + Placebo (Randomized)
Number analyzed (Participants) | 77 | 78
percentage of participants | 35.1 | 28.2
Statistical Analysis 1: Comparison: TCZ + MTX (Randomized) vs TCZ + Placebo (Randomized); Test type: Superiority or Other; p = 0.358, Chi-squared

5. Secondary Outcome: Change in the Health Assessment Questionnaire Disability Index (HAQ-DI) From Week 16 to Week 28
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0 = no difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Week 16 and Week 28
Population: ITT Population; only participants with non missing values were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ + MTX (Randomized) | TCZ + Placebo (Randomized)
Number analyzed (Participants) | 80 | 82
units on a scale | 0.08 (0.47) | 0.00 (0.52)
Statistical Analysis 1: Comparison: TCZ + MTX (Randomized) vs TCZ + Placebo (Randomized); Test type: Superiority or Other; p = 0.674, ANCOVA; Difference in Least Square (LS) Mean = 0.032, 95% CI 2-sided [-0.119 to 0.184] — Analysis of covariance (ANCOVA) model with treatment as factor and DAS28 value at Week 16 as covariate

6. Secondary Outcome: Change in the Quality of Life Questionnaire (Short Form-12 [SF-12]) From Week 16 to Week 28 in Mental Health
Description: Quality of life questionnaire (SF-12) scores were computed using the scores of 12 questions and ranged from 0 to 100, where a 0 score indicated the lowest level of health measured by the scales and 100 indicated the highest level of health. A negative change from baseline indicated decline in health and higher scores indicated improvement in health.
Time Frame: Week 16 and Week 28
Population: ITT Population; only participants with non missing values were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ + MTX (Randomized) | TCZ + Placebo (Randomized)
Number analyzed (Participants) | 79 | 79
units on a scale | -2.36 (10.22) | -0.38 (9.25)
Statistical Analysis 1: Comparison: TCZ + MTX (Randomized) vs TCZ + Placebo (Randomized); Test type: Superiority or Other; p = 0.204, ANCOVA; Difference in LS Mean = -1.873, 95% CI 2-sided [-4.775 to 1.030] — ANCOVA model with treatment as factor and mental component score (MCS) as covariate

7. Secondary Outcome: Change in the Quality of Life Questionnaire (SF-12) From Week 16 to Week 28 in Physical Health
Description: Quality of life questionnaire (SF-12) scores were computed using the scores of 12 questions and ranged from 0 to 100, where a 0 score indicated the lowest level of health measured by the scales and 100 indicated the highest level of health. A negative change from baseline indicated a worsening of quality of life.
Time Frame: Week 16 and Week 28
Population: ITT Population; only participants with non missing data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ + MTX (Randomized) | TCZ + Placebo (Randomized)
Number analyzed (Participants) | 79 | 79
units on a scale | 0.48 (9.49) | -2.26 (8.82)
Statistical Analysis 1: Comparison: TCZ + MTX (Randomized) vs TCZ + Placebo (Randomized); Test type: Superiority or Other; p = 0.015, ANCOVA; Difference in LS Mean = 3.376, 95% CI 2-sided [0.676 to 6.076] — ANCOVA model with treatment as factor and physical component score (PCS) as covariate

8. Secondary Outcome: Change From Week 16 to Week 28 in Global Assessment of Disease Activity as Assessed With the Visual Analogue Scale (VAS) Performed by Participant
Description: Participants were asked to rate their global assessment of disease activity on a scale ranging from 0=very good to 100=very bad. The scale was represented by a line with 0 at the left edge and 100 at the right edge. The participant was asked to mark the line corresponding to the assessment of their disease activity. The distance from the left edge was measured in mm.
Time Frame: Week 16 and Week 28
Population: ITT Population; only participants with non missing values were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ + MTX (Randomized) | Tocilizumab + Placebo (Randomized)
Number analyzed (Participants) | 82 | 82
units on a scale | 1.68 (23.80) | 0.56 (20.42)
Statistical Analysis 1: Comparison: TCZ + MTX (Randomized) vs Tocilizumab + Placebo (Randomized); Test type: Superiority or Other; p = 0.769, ANCOVA; Difference in LS Mean = 0.969, 95% CI 2-sided [-5.526 to 7.464] — ANCOVA model with treatment as factor and VAS performed by the participant at Week 16 as a covariate

9. Secondary Outcome: Change From Week 16 to Week 28 in Global Assessment of Disease Activity Assessed Using the VAS Performed by the Investigator
Description: as for outcome 8
Time Frame: Week 16 and Week 28
Population: ITT Population; only participants with non missing values were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ + MTX (Randomized) | TCZ + Placebo (Randomized)
Number analyzed (Participants) | 82 | 81
units on a scale | 2.71 (16.96) | 2.85 (18.48)
Statistical Analysis 1: Comparison: TCZ + MTX (Randomized) vs TCZ + Placebo (Randomized); Test type: Superiority or Other; p = 0.655, ANCOVA; Difference in LS Mean = -1.216, 95% CI 2-sided [-6.573 to 4.141] — ANCOVA model with treatment as factor and VAS performed by the investigator at Week 16 as covariate

ADVERSE EVENTS:
Time Frame: From Day 1 up to Week 36
Description: The data were planned per the protocol to be reported separately for pre-randomization period and post-randomization period.
Groups:
- TCZ + MTX (Pre-randomization): Participants received TCZ 8 mg/kg (maximum 800 mg) via IV infusion q4w up to Week 16 (total of 4 infusions). Participants also received MTX capsules, orally at a stable dose (10, 15, 17.5, or 20 mg/week but no maximum dose was set) weekly, up to Week 16. Participants with a response were randomized to receive TCZ and MTX in the second part of the study. Response was defined as participants having DAS28 score less than or equal to (<=)3.2.
- TCZ + Placebo (Pre-randomization): Participants received TCZ 8 mg/kg (maximum 800 mg) via IV infusion q4w up to Week 16 (total of 4 infusions). Participants also received MTX capsules, orally at a stable dose (10, 15, 17.5, or 20 mg/week but no maximum dose was set) weekly, up to Week 16. Participants with a response were randomized to receive TCZ and matching MTX placebo in the second part of the study. Response was defined as participants having DAS28 score <=3.2.
- TCZ + MTX (Post-randomization): TCZ 8 mg/kg (maximum 800 mg) q4w via IV infusion up to Week 16 (total of 4 infusions). Participants also received MTX capsules, orally, at a stable dose (10, 15, 17.5, or 20 mg/week but no maximum dose was set) weekly, up to Week 16. Participants with a response were randomized to receive 3 additional IV infusions of TCZ 8 mg/kg between Week 16 and Week 24 and MTX capsules, orally, at a stable dose (10, 15, 17.5, or 20 mg per week, but no maximum dose was set), weekly through Week 24. Response was defined as participants having DAS28 score <=3.2.
- TCZ + Placebo (Post-randomization): TCZ 8 mg/kg (maximum 800 mg) q4w via IV infusion up to Week 16 (total of 4 infusions). Participants also received MTX capsules, orally, at a stable dose (10, 15, 17.5, or 20 mg/week but no maximum dose was set) weekly, up to Week 16. Participants with a response were randomized to receive 3 additional IV infusions of TCZ 8 mg/kg between Week 16 and Week 24 and matching placebo MTX capsules, orally, at a stable dose (10, 15, 17.5, or 20 mg per week, but no maximum dose was set), weekly through Week 24. Response was defined as participants having DAS28 score <=3.2.
Arm/Group | TCZ + MTX (Not Randomized) | TCZ + MTX (Pre-randomization) | TCZ + Placebo (Pre-randomization) | TCZ + MTX (Post-randomization) | TCZ + Placebo (Post-randomization)
Serious Adverse Events (participants affected / at risk) | 11/96 | 0/83 | 1/82 | 1/83 | 4/82
Other Adverse Events (participants affected / at risk) | 28/96 | 20/83 | 24/82 | 8/83 | 4/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TCZ + MTX (Not Randomized) (N=96) | TCZ + MTX (Pre-randomization) (N=83) | TCZ + Placebo (Pre-randomization) (N=82) | TCZ + MTX (Post-randomization) (N=83) | TCZ + Placebo (Post-randomization) (N=82)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 3 | 0 | 0 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Salpingitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TCZ + MTX (Not Randomized) (N=96) | TCZ + MTX (Pre-randomization) (N=83) | TCZ + Placebo (Pre-randomization) (N=82) | TCZ + MTX (Post-randomization) (N=83) | TCZ + Placebo (Post-randomization) (N=82)
Leukopenia (Blood and lymphatic system disorders) | 7 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 3 | 6 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 15 | 12 | 10 | 8 | 4
Urinary tract infection (Infections and infestations) | 0 | 3 | 5 | 0 | 0
Respiratory tract infection (Infections and infestations) | 5 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 | 2 | 6 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.